CLINICAL TRIAL: NCT00004815
Title: Descriptive Study of Recombinant Human Insulin-Like Growth Factor for Osteoporosis in Werner's Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); University of Texas (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Non-Randomized | Purpose: Treatment
Other Study IDs: 199/12024; UTSMC-49215300
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-07

CONDITIONS: Werner's Syndrome
Keywords: Werner's syndrome; genetic diseases and dysmorphic syndromes; rare disease
MeSH Terms: conditions — Werner Syndrome; Genetic Diseases, Inborn; Rare Diseases | interventions — Growth Hormone

INTERVENTIONS:
Drug: growth hormone

SUMMARY:
OBJECTIVES:

I. Assess the safety and efficacy of recombinant human insulin-like growth factor 1 in a patient with Werner's syndrome and osteoporosis.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: The patient receives subcutaneous recombinant human insulin-like growth factor 1 daily for 7 months. The dose is adjusted according to the serum hormone level and biological markers of bone turnover.

Concurrent therapy includes a metabolic diet, calcium citrate, and estradiol.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Werner's syndrome with osteoporosis and low serum insulin-like growth factor 1 level Patient treated on protocol 04-9215300 "Metabolic and Skeletal Effects of Exogenous Recombinant Human Insulin-Like Growth Factor"

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1
Dates: Start 1992-05

CONTACTS AND LOCATIONS:
Overall Officials: Craig D. Rubin, Study Chair — University of Texas